CLINICAL TRIAL: NCT03481205
Title: Ischemic Conditioning During Air tRansport Save penUmbral Tissue
Acronym: ICARUS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Enrique Leira (Other)
Responsible Party: Sponsor-Investigator, Enrique Leira, Professor of Neurology, University of Iowa
Organization: University of Iowa (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 201712791
Record Dates: First submitted 2018-03-13; First posted 2018-03-29 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Acute Stroke
Keywords: remote limb ischemic conditioning; large vessel occlusion; helicopter transport
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Ischemic Conditioning (Experimental): Doctormate device used en route to the comprehensive stroke center
  Interventions: Device: Ischemic conditioning device

INTERVENTIONS:
Device: Ischemic conditioning device — RLIC will be done using a specialized blood pressure device ( Doctormate) that inflates to 200 mm HG for 5 minutes followed by 5 minutes deflation.
  Other Names: Standard medical care

SUMMARY:
The purpose of this study is to demonstrate the feasibility of performing remote limb ischemic conditioning (RLIC) using the Doctormate device, a special blood pressure device used to perform RLIC, on patients with acute ischemic stroke due to large vessel occlusion being transported to a thrombectomy capable center by the helicopter.

DETAILED DESCRIPTION:
In this study, 15 subjects presenting to a community hospital with signs and symptoms of ischemic stroke due to large vessel occlusion, transported to a comprehensive stroke center by aircew will receive RLIC using the Doctormate device.

The RLIC treatment will consist of 3-5 cycles ( depending on transportation time) of 5 minutes inflations of both blood pressure cuffs simultaneously. Blood pressure will be 200 mm HG with 5 minutes of reperfusion between each inflation.

Subjects will be evaluated upon arrival to the comprehensive stroke center and evaluated for side effects.

The study will be conducted at one site ( University of Iowa Hospitals and Clinics)

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 and ≤ 80 years
2. Suspected acute ischemic stroke with symptoms suggestive of large vessel occlusion (aphasia, agnosia, neglect, visual field cut, and gaze preference).
3. Patient screened for rtPA, and rtPA administered if eligible
4. Subject or legally authorized representative able to provide consent at the time of the assessment
5. NIHSS 6-20

Exclusion Criteria:

1. Any intracranial hemorrhage (parenchymal, subarachnoid, subdural, epidural) on CT scan at the community hospital
2. History of upper or lower extremity ischemia, known subclavian, brachial artery, iliac or femoral artery stenosis, subclavian steal syndrome, any upper or lower extremity soft tissue, orthopedic or vascular injury, or mastectomy or other procedure that may contraindicate taking blood pressure or having a cuff on the arm or leg for the conditioning treatment
3. History of diabetes mellitus
4. Enrollment in another clinical trial
5. Patient incarcerated
6. Pregnancy. Patients ages 18-55 will need to have a negative urine or blood based pregnancy test.
7. Agitation deemed unsafe for ischemic preconditioning testing.
8. Arteriovenous fistula in upper limb

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluate the feasibility of delivering RLIC by air medical crews in patients with AIS. This will be assessed by recording the number of cycles completed during transport. | The duration of the flight, typically 30 min-3 hours depending on weather and distance of the community hospital
  Feasibility will be assessed based on the number of cycles performed during transportation by air as follows:
  For flight time of duration of ≥ 60 minutes, ≥ 60% of subjects should receive 4 cycles of RLIC.
  For flight time of duration of 30-60 minutes, ≥ 60% of subjects should receive at least 3 cycles of RLIC.
  For flight duration of < 30 minutes, ≥60% of subjects should receive at least 2 cycle of RLIC.

SECONDARY OUTCOMES:
Assess adverse events related to performing RLIC in patients with large vessel occlusion. | AEs will be assessed during transport by aircrew, at 24 hours of admission and at 90 days.
  We will collect data on adverse events, severe and serious adverse events during transport, at 24 hours of hospital admission as well as at the 3 months follow up visit. An intendent medical monitor will be designated to evaluate the reported serious and related adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Enrique Leira, MD, Principal Investigator — University of Iowa Hospitals and Clinics- 200 Hawkins Dr, Iowa City, IA 52242
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No